CLINICAL TRIAL: NCT03099681
Title: Epithelioid Sarcoma. An Observational Study
Brief Title: An Observational Study on Epithelioid Sarcoma
Acronym: EPISObs
Status: Recruiting | Type: Observational
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Other Study IDs: ISG-EPISObs
Record Dates: First submitted 2017-03-17; First posted 2017-04-04 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Epithelioid Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor sample materiale
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Epitheloid Sarcoma patients: Patients with diagnosis of localized or advanced epitheloid sarcoma seen in the Italian reference centers for sarcoma treatment that receive treatment for Epitheloid Sarcoma
  Interventions: Other: Treatment for Epitheloid Sarcoma

INTERVENTIONS:
Other: Treatment for Epitheloid Sarcoma — Treatment Epitheloid Sarcoma according the disease guideline

SUMMARY:
Prospective Italian study aimed to provide a description of the population affected by Epithelioid Sarcoma (ES)

DETAILED DESCRIPTION:
The present prospective national study aims to provide a description of the population affected by ES, an insight into the natural history of the disease and an answer some on the outstanding questions on its management. Also, it will focus on enhancing any differences between the two ES variants (classical-type and proximal-type) in order gain a better understanding of the disease, tailor the treatment and lastly improve outcome.

ELIGIBILITY:
Inclusion criteria

1. Histological diagnosis of epithelioid sarcoma according to 2014 World Health Organization (WHO) classification, performed on biopsy or surgical specimen
2. Signed informed consent
3. Adequate patient compliance to treatment or follow up
4. No age limit

Exclusion criteria

1. Other malignancies within past 5 years, with exception of carcinoma in situ of the cervix and basocellular skin cancers treated with eradicating intent
2. Impossibility to ensure adequate compliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient affected by epithelioid sarcoma according to 2014 WHO classification
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-08-22 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Type of treatment given to patients with ES | From diagnosis until the date of death from any cause assessed up to 60 months
  Number of chemotherapy treatment received patients affected by ES

SECONDARY OUTCOMES:
Radiotherapy treatments | From the time of diagnosis and then every 6 months up to 60 months
  Number of patients affected by localized ES who received radiotherapy
Chemotherapy treatments | From the time of diagnosis and then every 6 months up to 60 months
  Number of patients affected by localized ES who received chemotherapy
Predictive biomarkers for response | At time of diagnosis and at the time of any progression where a biopsy is performed up to 60 months
  Tumor biomarkers expression in tumor tissue of patients affected by ES

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Casali, MD, Principal Investigator — Fondazione IRCCS INT Milano
Locations (11):
- Italy (11):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - IRST, Meldola, FC
  - Istituto Europeo di Oncologia, Milan, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Azienda Ospedaliera Universitaria Paolo Giaccone, Palermo, PA
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo, Torino
  - Istituto Ortopedico Rizzoli - Unit of Chemotherapy of Muscoloskeletal Tumors, Bologna
  - Fondazione IRCCS INT Milano, Milan
  - Irccs Istituto Oncologico Veneto (Iov), Padua
  - Ospedale Misericordia e Dolce Ist. Toscano Tumori, Az. USL4, Prato
  - Campus Biomedico, Roma
  - Istituti Fisioterapici Ospitalieri di Roma, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thway K, Jones RL, Noujaim J, Fisher C. Epithelioid Sarcoma: Diagnostic Features and Genetics. Adv Anat Pathol. 2016 Jan;23(1):41-9. doi: 10.1097/PAP.0000000000000102. PMID 26645461
- [Background] Guillou L, Wadden C, Coindre JM, Krausz T, Fletcher CD. "Proximal-type" epithelioid sarcoma, a distinctive aggressive neoplasm showing rhabdoid features. Clinicopathologic, immunohistochemical, and ultrastructural study of a series. Am J Surg Pathol. 1997 Feb;21(2):130-46. doi: 10.1097/00000478-199702000-00002. PMID 9042279
- [Background] Chase DR, Enzinger FM. Epithelioid sarcoma. Diagnosis, prognostic indicators, and treatment. Am J Surg Pathol. 1985 Apr;9(4):241-63. PMID 4014539
- [Background] Bos GD, Pritchard DJ, Reiman HM, Dobyns JH, Ilstrup DM, Landon GC. Epithelioid sarcoma. An analysis of fifty-one cases. J Bone Joint Surg Am. 1988 Jul;70(6):862-70. PMID 3392084
- [Background] Halling AC, Wollan PC, Pritchard DJ, Vlasak R, Nascimento AG. Epithelioid sarcoma: a clinicopathologic review of 55 cases. Mayo Clin Proc. 1996 Jul;71(7):636-42. doi: 10.1016/S0025-6196(11)63000-0. PMID 8656704